CLINICAL TRIAL: NCT04301089
Title: A Phase II Feasibility Trial Using Immersive Virtual Reality (VR) at the Time of Clinical Evaluation to Improve Psychological Distress and Anxiety in Primary Brain Tumor (PBT) Patients
Brief Title: Immersive Virtual Reality (VR) at the Time of Clinical Evaluation to Improve Psychological Distress and Anxiety in Primary Brain Tumor (PBT) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200065; 20-C-0065
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02-13

CONDITIONS: Anxiety
Keywords: Therapeutic VR Platform; Scanxiety; Brain Cancer; Brain Tumors
MeSH Terms: conditions — Anxiety Disorders; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental intervention (Experimental): Experimental VR Intervention, Survey or Questionnaire Completion and Sample Submission
  Interventions: Device: Pico G2 4K Headset with Applied VR software

INTERVENTIONS:
Device: Pico G2 4K Headset with Applied VR software — headset worn at time points defined in study

SUMMARY:
Background:

Distress, anxiety, and other psychological disorders may be more common in people with primary brain tumors (PBTs). PBTs can affect their symptoms, quality of life, and their tolerance of cancer treatments. Researchers want to learn if virtual reality (VR) technology can help reduce stress and improve mood. VR uses computer technology to make fake experiences and environments that look real. This allows people to escape from their lives and experience more positive thoughts and emotions.

Objective:

To learn if it is feasible to use a VR relaxation intervention in people with PBTs.

Eligibility:

Adults 18 and older who have a brain tumor and have recently reported psychological distress during their participation in the Natural History Study (NHS), protocol #16C0151

Design:

The VR intervention and all patient-reported outcome measures (PROs) will be done remotely using telehealth.

Participants will be mailed a VR headset. This headset looks like a thick pair of goggles that is worn over the eyes. Participants will view computer-generated environments on this VR headset.

Participants will fill out symptoms questionnaires at 4 different times points during participation in this study, including questionnaires for the NHS as well as 4 questionnaires unique to this study. There are also optional saliva samples collected at these timepoints. The 4 timepoints are:

* Before the VR intervention
* After the VR intervention
* 1 week later
* 4 weeks later

Participants will also have a phone interview 1 week after the initial VR interevention, which will last 10 to 15 minutes.

Participation lasts 4 to 6 weeks.

DETAILED DESCRIPTION:
Background

* Psychological distress is a common concern for patient across the cancer trajectory, which has been associated with worse clinical outcomes in terms of quality of life, adherence to treatment regimens, satisfaction with care, and poorer survival in past research.
* Virtual reality (VR) has the potential to alleviate some of the negative aspects of illness by allowing individuals to escape from their lives and experience more positive thoughts and emotions, which can be accomplished using cardiac coherence breathing techniques and distraction (both of which can improve psychological symptoms).
* Past VR research has shown promising improvements in anxiety, pain, distress and distraction through use of immersive VR interventions, though there is scant evidence in PBT populations, particularly in the time period surrounding their neuroimaging and clinical appointments when distress and anxiety can be highest.
* Recent evidence has demonstrated that the COVID-19 pandemic and associated mitigation procedures introduce additional stress for cancer patients, with higher levels of anxiety, depression, loneliness, and financial toxicity being reported during this time.
* The purpose of this phase II clinical trial is to determine the feasibility of implementing an immersive VR relaxation intervention in a PBT population and to assess the efficacy of the intervention to improve psychological distress and anxiety at the time of clinical evaluation. VR is an innovative delivery approach to teach our patients validated breathing and mindfulness techniques that can improve their psychological symptoms and their ability to self-manage these symptoms.

Objectives

-To describe the feasibility of implementing a VR intervention in a PBT population, including eligibility, accrual, compliance, adverse device effects, study completion, and participant satisfaction with the intervention

Eligibility

* PBT patients enrolled on the Natural History Study (NHS) trial in the Neuro-Oncology Branch (NOB) (all tumor types and grades eligible)
* Patients can be newly diagnosed, receiving active treatment, or on surveillance
* Adults (greater than or equal to 18 years of age) who are English-speaking and able to self-report symptoms
* Active corticosteroid therapy is permissible
* Exclude patients without tissue diagnosis, recent cranial surgery (less than or equal to 2 weeks), scalp wound healing issues, or seizures within the last 6 weeks
* Participants have reported greater than or equal to 1 on distres item from MDASI-BT prior to past clinic appointment
* Exclude patients who have a hypersensitivity to motion, severe nausea, or visual field deficits that might interfere with VR experience
* Exclude patients with a current diagnosis of generalized anxiety disorder (GAD), post-traumatic stress disorder (PTSD), claustrophobia, or panic disorder
* Those with visual deficits that might interfere with the VR experience, including hemianopsia, diplopia, and agnosia, based on their most recent clinical assessment

Design

* This is a phase II feasibility clinical trial with a single arm experimental design. The VR intervention and all patient-reported outcome measures (PROs) will be done remotely using telehealth.
* Study will include collection of self-reported PROs for distress, anxiety, mood disturbance, symptom burden/interference, quality of life, cognitive function, loneliness, and financial toxicity, as well as optional salivary stress biomarkers. These measures will be collected at baseline and immediately after a brief VR relaxation intervention to determine acute effects on distress, anxiety, and biological stress measures. Repeat post-intervention assessments will be done approximately 1 week and 1 month following the initial intervention to determine sub-acute effects on distress and anxiety, as well as impact on other symptoms. A semi-structured qualitative interview will also be conducted 1 month after the initial intervention to assess participant satisfaction with the intervention and how the pandemic has affected their psychological symptoms.
* Descriptive statistics, T-tests, Wilcoxon rank sum tests, and multiple logistic regression models will be used to evaluate the feasibility of the VR intervention. Linear mixed models and effect size calculations will be used to evaluate the acute and sub-acute effects of the VR intervention on self- reported PROs. Pearson or Spearman correlations will be used to evaluate the relationship between the biological stress measures and self-reported PROs.
* A total of 120 PBT patients will participate in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Primary brain tumor (PBT) patients enrolled on the Natural History Study (NHS) trial (16C0151) in the Neuro-Oncology Branch (NOB) who have an upcoming scan and clinical appointment
* Participants can be newly diagnosed, receiving active treatment, or on surveillance
* Concurrent enrollment in other NOB trials is permissible
* Adults (greater than or equal to 18 years of age) who are English-speaking
* Participants must be able to reliably self-report symptoms, based on clinician assessment
* Participants report greater than or equal to 1 on distress item from MDASI-BT prior to clinic appointment
* Active corticosteroid therapy is permissible
* Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Participants who do not have a tissue diagnosis (no past surgery or biopsy to confirm diagnosis)
* Cranial surgery less than or equal to 2 weeks prior to initiation of study intervention
* Scalp wound healing issues that might interfere with comfortable VR headset use
* Those who have epilepsy or have had a seizure in the last 6 weeks
* Participants with a current diagnosis of generalized anxiety disorder (GAD), post-traumatic stress disorder (PTSD), claustrophobia, or panic disorder
* Participants who have a hypersensitivity to motion or severe nausea, which could make the VR experience uncomfortable
* Those with visual deficits that might interfere with the VR experience, including hemianopsia, diplopia, and agnosia based on their most recent clinical assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete the sessions and questionnaires | End of Study
  To describe the feasibility of implementing a VR intervention in a PBT population, including eligibility, accrual, compliance, adverse events, study completion, and participant satisfaction with the intervention

SECONDARY OUTCOMES:
Measurement of mood disturbance | End of Study
  To assess the effects of a VR intervention on self-reported mood disturbance (as measured by PROMIS -Anxiety & PROMIS -Depression Short Forms) and symptom burden and interference (as measured by the MD Anderson Symptom Inventory Brain Tumor [MDASI-BT])
Measurement of distress and anxiety | End of Study
  To determine if the effects VR has on distress and anxiety are more pronounced in those with high distress (based on DT cut-off score of greater than or equal to 5) compared those with to low distress (based on DT scores of 0 4)
Measurement of Distress | End of Study
  To assess the effects of a VR intervention on self-reported acute and subacute distress (as measured by the NCCN Distress Thermometer [DT]) and anxiety (as measured by the State Anxiety Inventory [STAI-6]) in PBT patients
Measurement and comparison of distress and anxiety on those on systemic corticosteroids | End of Study
  To determine if the effects VR has on distress and anxiety are more pronounced in those individuals not on systemic corticosteroids (CS) compared to those who are

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L King, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
BTRIS: All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol = YES@@@@@@Statistical Analysis Plan (SAP) = YES@@@@@@Informed Consent Plan (ICF) = YES
Access Criteria: All studies due to BTRIS: Clinical data available during the study and indefinitely.

REFERENCES:
- [Background] Lin L, Chiang HH, Acquaye AA, Vera-Bolanos E, Gilbert MR, Armstrong TS. Uncertainty, mood states, and symptom distress in patients with primary brain tumors: analysis of a conceptual model using structural equation modeling. Cancer. 2013 Aug 1;119(15):2796-806. doi: 10.1002/cncr.28121. Epub 2013 May 9. PMID 23661311
- [Background] Maples-Keller JL, Bunnell BE, Kim SJ, Rothbaum BO. The Use of Virtual Reality Technology in the Treatment of Anxiety and Other Psychiatric Disorders. Harv Rev Psychiatry. 2017 May/Jun;25(3):103-113. doi: 10.1097/HRP.0000000000000138. PMID 28475502
- [Background] Niki K, Okamoto Y, Maeda I, Mori I, Ishii R, Matsuda Y, Takagi T, Uejima E. A Novel Palliative Care Approach Using Virtual Reality for Improving Various Symptoms of Terminal Cancer Patients: A Preliminary Prospective, Multicenter Study. J Palliat Med. 2019 Jun;22(6):702-707. doi: 10.1089/jpm.2018.0527. Epub 2019 Jan 24. PMID 30676847
- [Derived] King AL, Acquaye-Mallory AA, Vera E, Mendoza T, Reyes J, Stockdill ML, Gilbert MR, Armstrong TS. Feasibility and preliminary efficacy of a virtual reality intervention targeting distress and anxiety in primary brain tumor patients at the time of clinical evaluation: Study protocol for a phase 2 clinical trial. BMC Cancer. 2023 Mar 21;23(1):262. doi: 10.1186/s12885-023-10671-2. PMID 36944930
- [Derived] King AL, Roche KN, Leeper HE, Vera E, Mendoza T, Mentges K, Acquaye-Mallory AA, Adegbesan KA, Boris L, Burton E, Choi A, Grajkowska E, Kunst T, Levine J, Lollo N, Miller H, Panzer M, Penas-Prado M, Pillai V, Polskin L, Reyes J, Sahebjam S, Stockdill ML, Theeler BJ, Wu J, Gilbert MR, Armstrong TS. Feasibility of a virtual reality intervention targeting distress and anxiety symptoms in patients with primary brain tumors: Interim analysis of a phase 2 clinical trial. J Neurooncol. 2023 Mar;162(1):137-145. doi: 10.1007/s11060-023-04271-0. Epub 2023 Mar 8. PMID 36884201
- [Derived] King AL, Acquaye AA, Mendoza T, Reyes J, Stockdill M, Gilbert MR, Armstrong TS, Vera E. Feasibility and preliminary efficacy of a virtual reality intervention targeting distress and anxiety in primary brain tumor patients at the time of clinical evaluation: Study protocol for a phase 2 clinical trial. Res Sq [Preprint]. 2023 Feb 16:rs.3.rs-2521990. doi: 10.21203/rs.3.rs-2521990/v1. PMID 36865245
- [Derived] King AL, Roche KN, Leeper HE, Vera E, Mendoza T, Mentges K, Acquaye AA, Adegbesan K, Boris L, Burton E, Choi A, Grajkowska E, Kunst T, Levine J, Lollo N, Miller H, Panzer M, Penas-Prado M, Pillai V, Polskin L, Reyes J, Sahebjam S, Stockdill M, Theeler BJ, Wu J, Gilbert MR, Armstrong TS. Feasibility of a virtual reality intervention targeting distress and anxiety symptoms in patients with primary brain tumors: Interim analysis of a phase 2 clinical trial. Res Sq [Preprint]. 2023 Jan 31:rs.3.rs-2522094. doi: 10.21203/rs.3.rs-2522094/v1. PMID 36789426
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0065.html